CLINICAL TRIAL: NCT05376696
Title: Assessing Behavioural and Electrophysiological Effects of Reading Intervention in School-age Children With Dyslexia
Brief Title: Behavioural and Physiological Measures of Young Students With Dyslexia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Armando Bertone, Principal Investigator, Director, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Intervention & EEG
Record Dates: First submitted 2022-04-25; First posted 2022-05-17 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: EEG
Keywords: EEG; N400; reading intervention; reading disability; pre-post
MeSH Terms: conditions — Dyslexia | interventions — SET protein, human

STUDY DESIGN:
Intervention Model Description: In this study, the students will be randomized to either the treatment group to receive the proposed intervention (Set for Variability) or the active control arm. This group will receive current best practices reading. After randomization, each participant will stay in their assigned treatment arm for ten weeks.
Who Masked: Participant
Masking Description: Students will not be told whether they are receiving the intervention or the active control treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Set for Variability (Experimental): Students in the experimental group will receive an average of 10-12 hrs. of small group intervention. All lessons will include (i) a focus on blending and segmenting phonemes within a synthetic phonics model, (ii) teaching common, vocabulary words (iii)shared book reading, and (iv) Set-for-variability component (SfV). This component will focus on teaching students how to find the sound variation of a grapheme-phoneme rule. For example when to use the sound /k/in /ch/ to read words such as "stomach"
  Interventions: Behavioral: Set For Variability
- Current best practices (Active Comparator): The control group will receive current-best practices (CBP). The participants will receive a similar approach as in the intervention group without Set-for-Variability. The participants will receive (i) a focus on blending and segmenting phonemes within a synthetic phonics model, (ii) vocabulary, (iii) shared book reading, and (iv) the absence of teaching Set-for-Variability. Instead of Set-for-variability, the participants will receive sight word reading of frequent words. They will learn the most frequent pronunciation of vowels: ee, ea, oo, ou, oa, ai, ay
  Interventions: Behavioral: Current Best Practices

INTERVENTIONS:
Behavioral: Set For Variability — This intervention will focus on training students to use a sound variation of grapheme correspondence rule in order to read an irregular spelling word correctly.
  Arms: Set for Variability
Behavioral: Current Best Practices — This active control intervention will focus on training students to use grapheme-phoneme correspondence rules and sight words in the absence of set-for-variability component
  Arms: Current best practices

SUMMARY:
The proposed is reading intervention study to track neural changes in the brain. Students with dyslexia will participate in a reading study. Pre and post-analysis data will be obtained to see whether there will be positive neural and behavioural change.

DETAILED DESCRIPTION:
A learning disability in reading is one of the most common neurobiological diagnoses in school-aged children. Statistics Canada reported that 3.2% of children in Canada have a learning disability (LD), making LD the most prevalent type of childhood condition. The new definition of LD has become more complicated to diagnose and treat children. Canadian universities invested recently in conducting research that tracks neural changes in the identification and remediation of LD. Electroencephalography (EEG) is one of the most common tools to inquire about brain information processing and neural changes. However, only one German study has used a reading intervention and EEG to track neural changes of children with LD in reading. This study delivered two reading interventions but did not report which intervention affected reading improvement. Hence, little is known about reading interventions that would induce positive neural changes in young children with LD. This proposal aims to implement a specific reading intervention in children and track neuronal changes. The results of this proposal will be invaluable in improving the predictive tools we use for early diagnosis of LD in reading, identifying better-targeted reading interventions, and in better allocation of resources to health and educational services.

To understand how the brain processes language in real-time, Event-Related Potential (ERPs) studies have been commonly used to assess the neural underpinnings of reading disability (RD), especially in children. Of particular interest, the N400 is a negative ERP waveform peaking at 400 milliseconds that is sensitive to the lexico-semantic aspect of language. The N400 represents an important language-relevant measure that can be used to investigate the neural basis of reading comprehension acquisition in typical readers, a process critical to reading development in school-age populations. The N400 assesses lexical-semantic processing when a student is introduced to a sentence with a pseudoword or a semantically incorrect word, as in "the pizza was too hot to cry." The N400 is sensitive in typical readers, indicating that they understand the semantic incongruity. There is also evidence that the N400 is atypical in individuals with reading disabilities and reading comprehension deficits.

These brain-based explanations give educational practice and understanding of the neural processes underlying reading difficulties, reading comprehension deficits, and potentially effective intervention mechanisms. Several studies demonstrate the potential relevance of neuroimaging for identifying a reading disability. Researchers have also shown that neural changes occur after a successful reading intervention. However, it remains unknown whether a reading intervention modulates reading-relevant brain activity, such as that of the N400.

One common approach to this problem is to teach common exception words by sight. An alternative approach some researchers have proposed is that in addition to teaching phonics, children are to be trained to "generate alternative pronunciations when they come to unknown words until they produce a pronunciation that is a real word, and which makes sense in context". This process is known as Set-for-Variability (SfV). For example, a child is taught the standard pronunciation of "ch" in the match, hatch, and catch. The child would then use this regularized pronunciation of "ch" to read the word stomach, an irregular spelled word. If a child fails to read the irregularly spelled word stomach using regularized pronunciation, then "the child has to change one or more sound associations and try again". Set-for-Variability is "the ability to determine the correct pronunciation of proximation to spoken English words". This means making a link from 'spelling pronunciations' (the product of synthetic phonics such as 'c'-'a'-'t' from the printed word 'cat') to a conventional pronunciation of that word. If pronouncing a word does not produce a meaningful phrase in context, the individual would need to try a different pronunciation.

The proposed study is a randomized-control study where thirty-eight students aged 6-7 years with a reading disability will be randomly assigned into a control and intervention group. The participants will be matched on age, IQ, and reading level before randomization. Participants in the control group will be included in a Current Best Practices (CBP) group and exposed to an intervention that focuses on grapheme-phoneme correspondence rules. In addition to the CBP, participants in the intervention group will receive 8-10 weeks of the Set-for-Variability intervention. Pre-post behavioural measures will be conducted to see if the Set-for-Variability intervention impacts word reading measured using validated assessment tools and the N400 amplitude. The present research will provide the first empirical data on the neural changes following a "Set-for-Variability"-based reading intervention.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis with Dyslexia from school psychologists, a psychiatrist

Exclusion Criteria:

* Have a comorbid diagnosis with ADHD and Autism
* Have Epilespy

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Physiological parameter using EEG | 10 weeks after baseline
  Time to detect the N400 after the onset of the target word at a window of 350-650 milliseconds. If the time of the N400 does not occur within this time frame window, this might indicate semantic integration deficits/and participant did not respond well to the intervention.

SECONDARY OUTCOMES:
Standardized reading measures | 10 weeks after baseline
  Reading measures: Castle and Coltheart Word reading, Woodcock Johnson grapheme phoneme, WIAT reading comprehension and Set-for-Variability. [Percentile range]. Scores between 75-97 percentile are considered average to above average. Scores between 9-25 percentile are considered low and below average. Depending on where the participant scores will show improvement or no improvement to the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kutas M, Federmeier KD. Thirty years and counting: finding meaning in the N400 component of the event-related brain potential (ERP). Annu Rev Psychol. 2011;62:621-47. doi: 10.1146/annurev.psych.093008.131123. PMID 20809790
- [Background] Hasko S, Groth K, Bruder J, Bartling J, Schulte-Korne G. What does the brain of children with developmental dyslexia tell us about reading improvement? ERP evidence from an intervention study. Front Hum Neurosci. 2014 Jun 26;8:441. doi: 10.3389/fnhum.2014.00441. eCollection 2014. PMID 25018723
- [Background] Tunmer WE, Chapman JW. The simple view of reading redux: vocabulary knowledge and the independent components hypothesis. J Learn Disabil. 2012 Sep-Oct;45(5):453-66. doi: 10.1177/0022219411432685. Epub 2012 Jan 31. PMID 22293683
- [Background] Schulz E, Maurer U, van der Mark S, Bucher K, Brem S, Martin E, Brandeis D. Impaired semantic processing during sentence reading in children with dyslexia: combined fMRI and ERP evidence. Neuroimage. 2008 May 15;41(1):153-68. doi: 10.1016/j.neuroimage.2008.02.012. Epub 2008 Mar 10. PMID 18378166
- See also: Castle and Coltheart grapheme-phoneme reading test — https://researchers.mq.edu.au/en/publications/the-castles-and-coltheart-test-2-cc2
- See also: Woodcock Johnson reading achievement test — https://www.hmhco.com/~/media/sites/home/hmh-assessments/clinical/woodcock-johnson/pdf/wjiii/wjiii_asb8.pdf?la=en
- See also: WIAT reading comprehension test — https://www.child-psychologist.com.au/wechsler-individual-achievement-test.html